CLINICAL TRIAL: NCT00869037
Title: Analgesia After Total Knee Arthroplasty: Randomized Controlled Trial Comparing (a) Periarticular Multimodal Technique With (B) Continuous Femoral Nerve Block + Posterior Capsular Injection
Brief Title: Analgesia After Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sanjay Aragola, Department of Anesthesia, Concordia General Hospital, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2008:123
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2010-01

CONDITIONS: Analgesia
Keywords: Randomized controlled study; Total knee arthroplasty; Post operative pain; Continuous Femoral Nerve Block; Posterior Capsular injection; Periarticular injection
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Periarticluar Multimodal Technique (Active Comparator)
  Interventions: Drug: Periarticular Injection
- CFNB plus Posterior Capsular Injection (Active Comparator)
  Interventions: Drug: CFNB + Posterior Capsular Injection

INTERVENTIONS:
Drug: Periarticular Injection — A 20 ml bolus of saline will be given through the sham femoral nerve block catheter. Periarticular infiltration solution containing 400 mg Ropivicaine, 30 mg Ketorolac, 5 mg Epidural Grade Morphine, and 0.6 ml of 1:1000 Epinephrine will be made up to a volume of 100 ml with saline. Intra-op, 20 ml will be injected into the posterior capsule; 40 ml in the quadriceps mechanism, retinacular tissues, medial and lateral collateral ligaments; 40 ml in the skin and subcutaneous tissues. The sham catheter will be connected to a saline infusion running at 15 ml/hr until the morning of post-operative day 2.
  Arms: Periarticluar Multimodal Technique
Drug: CFNB + Posterior Capsular Injection — A 20 ml bolus of 0.2% Ropivacaine will be given via a femoral nerve catheter. Periarticular infiltration will be performed intra-op. 20 ml of 1% Ropivacaine in the posterior capsule; 20 ml of normal saline in the quadriceps mechanism, retinacular tissues, medial and lateral collateral ligaments; 20 ml of normal saline for the skin and subcutaneous tissues. Postoperatively, the femoral catheter will be infused with 0.15% Ropivacaine running at 15 ml/hour until the morning of post-operative day 2
  Arms: CFNB plus Posterior Capsular Injection

SUMMARY:
The recovery from knee replacement surgery often involves a significant amount of pain. The best way to prevent/treat this pain is unknown. This study will compare two accepted methods of pain control in order to determine which is superior. The first method involves the injection of a solution containing multiple medications into the knee joint at the time of surgery. The second method involves the placement of a catheter adjacent to the femoral nerve which senses pain from the knee. This catheter is used to deliver local anesthetic which serves to block the transmission of pain signals from the nerve. The catheter will be left in place until 2 days after surgery. This method is combined with injection of local anesthetic in a particular area of the knee joint at the time of surgery. Patients will be followed until 2 days after surgery in order to determine which method is superior. We believe the second method will be deemed superior.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II, & III patients
* Elective primary total knee arthroplasty
* Spinal Anesthesia

Exclusion Criteria:

* Patients refusing consent
* Contraindications to regional anesthesia
* Pre-existing neurological disease
* Allergy/contraindication to drugs used in the study
* Revision knee arthroplasty
* Patients with chronic pain/on narcotics preoperatively
* Pre-existing Rheumatoid Arthritis/Ankylosing Spondylitis
* Alcohol or drug abuse
* Psychiatric disorders
* Inability to use the outcome assessment tools
* Wheel chair or walker dependent for mobilization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-07 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Static and dynamic pain scores until post-operative day 2 (POD 2) | 9:00 and 15:30 daily for the first 2 postoperative days

SECONDARY OUTCOMES:
Equivalent narcotic consumption until POD 2 | 9:00 and 15:30 daily until POD 2
Number of patients requiring Ketamine and ketamine dosage for intractable pain | 9:00 and 15:30 daily until POD 2
Number of patients requiring Cryo-Cuff for intractable pain | 9:00 and 15:30 daily until POD 2
Number of patients with pain scores in the mild (numerical rating scale 0-3), moderate (NRS 3-7) and severe (NRS 7-10) range | 9:00 and 15:30 daily until POD 2
Incidence of narcotic related side effects (nausea, vomiting, pruritis, euphoria, dysphoria, hallucination, respiratory depression) | 9:00 and 15:30 daily until POD 2
Number of patients able to mobilize with or without a frame | POD 1-2
Maximum knee flexion (active/passive) | POD 1-2, at discharge, and at first follow-up visit
Hospital length of stay | Until Hospital discharge
Patient satisfaction scores | POD 0-2, at hospital discharge, and at first postoperative follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Aragola, MD, FRCA, Principal Investigator — University of Manitoba; Marshall S Tenenbein, MD, Principal Investigator — University of Manitoba
Locations (1):
- Concordia Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Aragola S, Arenson B, Tenenbein M, Bohm E, Jacobsohn E, Turgeon T. Prospective randomized trial of continuous femoral nerve block with posterior capsular injection versus periarticular injection for analgesia in primary total knee arthroplasty. Can J Surg. 2021 Apr 28;64(3):E265-E272. doi: 10.1503/cjs.020519. PMID 33908425